CLINICAL TRIAL: NCT00310206
Title: A Randomized, Open-Label, Phase I Clinical Trial Comparing the Safety, Reactogenicity, and Immunogenicity of Immunization With Inactivated Influenza A/H5N1 Vaccine Administered by the Intradermal or the Intramuscular Route Among Healthy Adults
Brief Title: H5N1 Vaccine Intramuscular Versus Intradermal in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 05-0015
Record Dates: First submitted 2006-03-30; First posted 2006-04-03 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2009-10

CONDITIONS: Influenza
Keywords: Influenza, pandemic, H5N1, vaccine
MeSH Terms: conditions — Influenza, Human; Influenza in Birds

ARMS (4):
- ID injection-9 mcg (Experimental): 25 subjects to receive 9 mcg of inactivated influenza A/H5N1 vaccine intradermally on Days 0 and 28.
  Interventions: Biological: Inactivated Influenza A Vaccine A/H5N1
- IM injection-15 mcg (Experimental): 25 subjects to receive 15 mcg of inactivated influenza A/H5N1 vaccine intramuscularly on Days 0 and 28.
  Interventions: Biological: Inactivated Influenza A Vaccine A/H5N1
- IM injection-45 mcg (Experimental): 25 subjects to receive 45 mcg of inactivated influenza A/H5N1 vaccine intramuscularly on Days 0 and 28.
  Interventions: Biological: Inactivated Influenza A Vaccine A/H5N1
- ID injection-3 mcg (Experimental): 25 subjects to receive 3 mcg of inactivated influenza A/H5N1 vaccine intradermally on Days 0 and 28.
  Interventions: Biological: Inactivated Influenza A Vaccine A/H5N1

INTERVENTIONS:
Biological: Inactivated Influenza A Vaccine A/H5N1 — Monovalent subvirion H5 vaccine (HA of A/Vietnam/1203/04), inactivated A/H5N1 vaccine administered intradermally (ID); doses: 3 or 9 micrograms.
  Arms: ID injection-3 mcg; ID injection-9 mcg
Biological: Inactivated Influenza A Vaccine A/H5N1 — Monovalent subvirion H5 vaccine (HA of A/Vietnam/1203/04), inactivated A/H5N1 vaccine administered intramuscularly (IM); doses: 15 or 45 micrograms.
  Arms: IM injection-15 mcg; IM injection-45 mcg

SUMMARY:
The purpose of this research study is to compare how the body reacts to different strengths of an H5N1 flu vaccine when given by different routes of injection (injection into the skin or into the muscle). It will also compare how antibodies (proteins produced by the body's immune system that recognize and help fight infections and other foreign substances in the body) are made after receiving the H5N1 flu vaccine. Participants will include 100 healthy adults, ages 18-40 years. Study procedures include blood samples and completing a memory aid documenting daily oral temperature and side effects for 7 days following each vaccination. Participants may be involved in the study for up to 13 months.

DETAILED DESCRIPTION:
This is a single-center, randomized, open-label, dose-ranging, phase I comparative trial of intradermal (ID) and intramuscular (IM) injection with subvirion inactivated influenza A/H5N1 vaccine in healthy adults, 18 to 40 years old, inclusive. This study is designed to investigate the safety, reactogenicity, and dose-related immunogenicity of an investigational inactivated influenza A/H5N1 virus vaccine given by ID injection compared to IM injection. The primary objectives of this study are to: compare dose-related safety and reactogenicity profiles of ID and IM injection with subvirion inactivated influenza A/H5N1 vaccine among healthy young adults; compare the dose-related immunogenicity of subvirion inactivated influenza A/H5N1 vaccine given by ID with vaccine given by IM injection among healthy young adults 1 month after receipt of the second dose of vaccine; and provide information for the selection of the best dose levels for further studies. The secondary objectives of this study are to: evaluate dose-related immunogenicity and the percent of subjects responding approximately 1 and 7 months after the first vaccination; and evaluate the dose-related safety, reactogenicity and immunogenicity following receipt of a third dose of vaccine administered 6-7 months after the second dose of vaccine. The study will have 2 comparison arms (IM and ID), and 2 dosage levels will be evaluated in each arm (4 vaccine groups total). Subjects will be randomized 1:1:1:1 (25 subjects in each group) to receive 2 doses 1 month apart of an inactivated influenza A/H5N1 vaccine containing 15 mcg or 45 mcg of H5 HA by the IM route; or one-fifth of the IM dose (3 mcg or 9 mcg) by the ID route. Subjects will maintain a memory aid recording oral temperature, and systemic and local adverse events for 7 days after each inoculation. Serum for immunogenicity evaluations will be obtained prior to first vaccination, at Day 0, prior to second vaccination, at Day 28, and on Day 56 and approximately Day 215 (7 months) after dose 1. This study is linked to DMID protocol 07-0022.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female (as indicated by a negative urine pregnancy test immediately prior to vaccine administration) between the ages of 18 and 40 years, inclusive.
* Women of childbearing potential who are at risk of becoming pregnant must agree to practice adequate contraception (i.e., barrier method, abstinence, and licensed hormonal methods) for at least 3 months after receipt of dose 2 (or dose 3, if applicable).
* Is in good health, as determined by vital signs (heart rate, blood pressure, oral temperature), medical history and a targeted physical examination based on medical history.
* Able to understand and comply with planned study procedures.
* Provides informed consent prior to any study procedures and is available for all study visits.
* Is not receiving any regular medications with the exceptions of birth control pills and vitamins.
* Meets all other inclusion criteria and must have received two doses of inactivated influenza A/H5N1 vaccine in the present study to be eligible for a third dose.

Exclusion Criteria:

* Has a known allergy to eggs or other components of the vaccine.
* Has a positive urine pregnancy test prior to vaccination (if female of childbearing potential), is lactating, or has the intention to become pregnant within 3 months of receipt of their second dose of vaccine.
* Is undergoing immunosuppression as a result of an underlying illness or treatment.
* Has an active neoplastic disease or a history of any hematologic malignancy.
* Is using oral or parenteral steroids, high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) or other immunosuppressive or cytotoxic drugs.
* Has a history of receiving immunoglobulin or other blood product within the 3 months prior to enrollment in this study.
* Has received any other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrollment in this study.
* Has an acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe or would interfere with the evaluation of responses (this includes, but is not limited to: known chronic liver disease, significant renal disease, unstable or progressive neurological disorders, diabetes mellitus, and transplant recipients).
* Has a history of severe reactions following immunization with contemporary influenza virus vaccines.
* Has an acute illness, including an oral temperature greater than 100.4 degrees Fahrenheit, within 1 week of vaccination.
* Received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to each vaccination in the study, or expects to receive an experimental agent within 1 month after each vaccination in the study.
* Prior receipt of influenza A/H5N1 vaccine, other than the present study.
* Is enrolled or planning to enroll in another interventional trial at any time between receipt of the third dose of vaccine and the end of the study (approximately 6 months after receipt of the third dose).
* Has any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2005-07; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects in each vaccine group achieving a serum neutralizing antibody titer of 1:40 against the influenza A/H5N1 virus. | Day 56.
Geometric mean titer (GMT) and proportion of subjects achieving a 4-fold or greater increase in serum neutralizing or hemagglutination inhibition (HAI) antibody titer in each group. | Day 56.
Adverse event (AE) or serious adverse event (SAE) information (solicited in-clinic and via memory aids and periodic targeted physical assessments). | Duration of study.

SECONDARY OUTCOMES:
Geometric mean titer (GMT) and proportion of subjects achieving a 4-fold or greater increase in neutralizing antibody titers in each group 1 and 7 months after receipt of dose 1. | Blood samples for serum assays will be collected prior to first dose on day 0, prior to second dose on day 28, and on days 56 and 215 after the first immunization.
GMT and the proportion of subjects achieving a 4-fold or greater increase in HAI and neutralizing antibody titers in each group 1 month after receipt of a 3rd dose of vaccine administered approximately 6-7 months after the 2nd dose of vaccine. | Blood samples for serum assays will be collected prior to first dose on day 0, prior to second dose on day 28, and on days 56 and 215 after the first immunization.
Development of serum antibody responses against antigenically drifted variants of H5 influenza virus. | Blood samples for serum assays will be collected prior to first dose on day 0, prior to second dose on day 28, and on days 56 and 215 after the first immunization.
Geometric mean titer (GMT) and proportion of subjects achieving a 4-fold or greater increase in HAI and neutralizing antibody titers in each group 1 and 7 months after receipt of dose 1. | Blood samples for serum assays will be collected prior to first dose on day 0, prior to second dose on day 28, and on days 56 and 215 after the first immunization.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States